CLINICAL TRIAL: NCT07336277
Title: Sleep Quality and the Efficacy of a Multimodal Sleep Pathway in Hospitalized Orthopedic Trauma Patients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: AO North America (Other)
Responsible Party: Principal Investigator, Mara Schenker, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2025P012693
Record Dates: First submitted 2026-01-07; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Orthopedic Trauma; Sleep Quality
Keywords: Multimodal Sleep Pathway; Sleep Quality; Opioid consumption
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Zolpidem; Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Multimodal Sleep Pathway (Experimental): Participants receive a multimodal sleep pathway consisting of pharmacologic sleep aids and non-pharmacologic sleep hygiene education beginning on the first postoperative night and continuing daily until hospital discharge.
  Interventions: Drug: Zolpidem; Dietary Supplement: Melatonin; Behavioral: Sleep Hygiene Education; Device: Actigraph GT3X-BT Actigraph
- Standard Care (Other): Participants receive routine postoperative care without sleep-specific pharmacologic or behavioral interventions. Standard pain management is provided per the clinical team's discretion.
  Interventions: Other: Standard Postoperative Care; Device: Actigraph GT3X-BT Actigraph

INTERVENTIONS:
Other: Standard Postoperative Care — Includes routine pain management and nursing care
  Arms: Standard Care
Drug: Zolpidem — * Dose: 5 mg
  * Administration: Taken nightly at bedtime
  * Purpose: Supports sleep initiation as part of the multimodal sleep pathway
  * Additional Notes: FDA-approved sedative-hypnotic used short-term for insomnia
  Arms: Multimodal Sleep Pathway
Dietary Supplement: Melatonin — * Dose: 3 mg
  * Administration: Taken 30 minutes before bedtime
  * Purpose: Supports circadian regulation and sleep continuity
  Arms: Multimodal Sleep Pathway
Behavioral: Sleep Hygiene Education — * Components: Guidance on consistent sleep schedules, minimizing nighttime disruptions, reducing screen exposure before bed, and optimizing environmental factors (light, noise, temperature)
  * Delivery: Provided by research staff daily during hospitalization
  Arms: Multimodal Sleep Pathway
Device: Actigraph GT3X-BT Actigraph — The ActiGraph GT3X-BT (ActiGraph, LLC; Pensacola, FL) is a lightweight, wrist-worn accelerometer used to objectively measure sleep-wake patterns in hospitalized patients. The device continuously records movement data that are processed using validated algorithms to estimate total sleep time, sleep efficiency, and number of awakenings.

SUMMARY:
The goal of this study is to determine whether a multimodal sleep pathway can enhance sleep quality in hospitalized patients with orthopedic trauma. It will also evaluate the effect of this pathway on opioid use and pain perception during recovery.

The main study questions are:

* Does the multimodal sleep pathway improve sleep quality and duration?
* Does the pathway reduce the amount of opioids patients use during hospitalization?
* Does improved sleep reduce pain interference with daily activities?

Researchers will compare the multimodal sleep pathway to standard postoperative care to see if the pathway helps patients sleep better and rely less on opioids.

Participants will:

* Receive either the multimodal sleep pathway (zolpidem, melatonin, and sleep hygiene education) or standard care
* Wear a wrist-worn actigraphy device to track sleep during their hospital stay
* Complete daily questionnaires about sleep quality and pain

DETAILED DESCRIPTION:
Post-surgical orthopedic trauma patients frequently experience significant sleep disturbances, including reduced sleep quality, increased nighttime awakenings, and shortened sleep duration. Sleep and pain have a bidirectional relationship in which poor sleep increases pain sensitivity, and higher pain levels further disrupt sleep. Experimental sleep-restriction studies have shown that pain perception increases after only two nights of partial sleep deprivation and continues to worsen with each additional night. Despite these established interactions, objective sleep metrics have not been well characterized in the orthopedic trauma inpatient population, where postoperative pain, environmental disruptions, and medication use may all contribute to sleep disturbance.

Sleep patterns are also influenced by psychoactive substances, including opioids. Substance use and sleep-wake regulation share overlapping neurobiological pathways, and disruptions in circadian rhythms can occur during substance use, withdrawal, or detoxification. Although the mechanisms by which opioids alter sleep architecture are not fully understood, prior studies have shown that opioid exposure reduces restorative sleep stages, including deep sleep and rapid eye movement (REM) sleep, while increasing lighter stage-2 sleep. These changes may contribute to fragmented sleep and impaired recovery in postoperative patients who rely on opioids for pain management.

Non-opioid strategies have shown promise in improving sleep quality in hospitalized and postoperative patient populations. Behavioral approaches such as relaxation techniques, stimulus control, and structured sleep hygiene have been associated with improvements in sleep duration and continuity. Pharmacologic alternatives, including zolpidem and melatonin, have demonstrated benefit in orthopedic and general adult populations by supporting sleep initiation, circadian regulation, and overall sleep quality.

This study builds on these findings through two complementary aims. Aim 1 analyzes previously collected actigraphy and survey data from a randomized controlled trial of adults with isolated orthopedic injuries (NCT04154384). In that study, participants wore wrist-worn actigraphy devices during hospitalization and completed validated sleep and pain assessments at baseline and postoperative follow-up visits. Preliminary analyses indicate that patients experience short, fragmented sleep and that higher opioid utilization may be associated with decreased sleep quantity and quality. Further analysis is needed to characterize these relationships using objective sleep metrics and detailed opioid timing and dosing data.

Aim 2 evaluates a multimodal sleep pathway designed to improve sleep quality and reduce opioid use during inpatient recovery. In a prospective randomized controlled trial, participants are assigned to receive either standard postoperative care or a sleep pathway that includes low-dose zolpidem, melatonin, and structured sleep hygiene education. The intervention begins on the first postoperative night and continues daily until discharge. Sleep outcomes are assessed using daily subjective questionnaires and continuous wrist actigraphy. Opioid consumption is recorded and converted to morphine milligram equivalents to allow standardized comparison. Pain perception is measured using validated patient-reported tools. Feasibility outcomes include recruitment, adherence to the intervention, actigraphy wear compliance, and retention through discharge. Safety monitoring includes assessment for medication-related side effects and actigraphy-related discomfort.

Together, these aims will provide foundational data on the relationship between opioid use and sleep quality in orthopedic trauma patients and will evaluate whether a structured multimodal sleep intervention can improve sleep and reduce reliance on opioids during hospitalization. Findings will inform the design of future larger-scale trials aimed at optimizing sleep and recovery in this population.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized with an isolated lower extremity orthopedic injury requiring surgical intervention.
* Expected hospital stay of at least 3 days.
* No known pre-existing sleep disorders.
* No current use of sleep aids, such as zolpidem or melatonin, before hospitalization

Exclusion Criteria:

* Participants with a history of chronic opioid use prior to hospitalization.
* Pre-existing diagnosed sleep disorders (e.g., obstructive sleep apnea, insomnia).
* Contraindications to zolpidem or melatonin use (e.g., allergies, interactions with other medications).
* Cognitive impairment or inability to comply with study procedures.
* Severe traumatic brain injury or other neurological conditions that may affect sleep or pain perception.
* Participants receiving mechanical ventilation or sedatives that significantly affect sleep architecture.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Total Sleep Time | Daily during inpatient hospitalization (approximately 3-7 days)
  Total minutes of sleep obtained each night, measured continuously using a wrist-worn actigraphy device (Actigraph GT3X-BT).
  Between-group differences in total sleep time will be evaluated using independent t-tests or Mann-Whitney U tests, depending on distribution. Longitudinal changes will be analyzed using linear mixed-effects models with random intercepts to account for repeated measures. Covariates may include age, injury characteristics, and baseline pain levels.
Sleep Efficiency | Daily during inpatient hospitalization (approximately 3-7 days)
  Percentage of time spent asleep while in bed, calculated from actigraphy data collected continuously during hospitalization.
  Group comparisons will be conducted using independent t-tests or nonparametric equivalents. Mixed-effects modeling will assess within-subject changes over time and the effect of group assignment.
Number of Awakenings | Daily during inpatient hospitalization (approximately 3-7 days)
  Total number of nighttime awakenings detected by actigraphy, reflecting sleep fragmentation.
  Awakening counts will be compared between groups using Poisson or negative binomial regression models, depending on dispersion. Mixed-effects count models will evaluate changes over time.
Subjective Sleep Quality: PROMIS scale | Daily during inpatient hospitalization (approximately 3-7 days)
  The PROMIS Sleep Disturbance Short Form assesses self-reported perceptions of sleep quality, sleep depth, and restoration over the past 7 days. Items are rated on 5-point Likert scales and summed to produce a raw score, which is converted to a standardized PROMIS T-score. Higher T-scores indicate greater sleep disturbance (worse sleep), and lower T-scores indicate less sleep disturbance (better sleep).
Subjective Sleep Quality: Leeds Sleep Evaluation Questionnaire (LSEQ) | Daily during inpatient hospitalization (approximately 3-7 days)
  The LSEQ is a 10-item patient-reported questionnaire that assesses subjective changes in sleep and early-morning functioning using 100-mm visual analogue scales. Items evaluate four domains: Getting to Sleep (GTS), Quality of Sleep (QOS), Awakening From Sleep (AFS), and Behavior Following Waking (BFW). Each item is scored from 0-100 mm, with higher scores indicating greater improvement relative to usual sleep and lower scores indicating worsening.
Daily Opioid Utilization | Daily during inpatient hospitalization (approximately 3-7 days)
  Total opioid consumption recorded from the medical record and converted to morphine milligram equivalents (MMEs) to allow standardized comparison across medication types and dosing regimens.

SECONDARY OUTCOMES:
Pain Interference | Daily during inpatient hospitalization (approximately 3-7 days)
  Patient-reported pain interference with daily activities measured using a validated pain interference scale. Higher scores indicate greater interference
Recruitment Feasibility | Throughout the study (upto 7 days of hospital stay)
  Assesses the proportion of eligible orthopedic trauma patients who enroll in the study during the inpatient recruitment window. Recruitment feasibility reflects the practicality of identifying, approaching, and enrolling participants in an acute trauma setting.
  Recruitment rate will be calculated as the number of enrolled participants divided by the number of eligible patients approached. Results will be summarized using proportions and 95% confidence intervals.
Adherence to Pharmacologic Components | Throughout the study (upto 7 days of hospital stay)
  Assesses adherence to the medication components of the multimodal sleep pathway, defined as the proportion of nights during which participants receive the prescribed low-dose zolpidem and melatonin as ordered.
  Adherence will be summarized as the percentage of scheduled doses administered. Means, standard deviations, and proportions will be reported.
Adherence to Non-Pharmacologic Components | Throughout the study (upto 7 days of hospital stay)
  Assesses adherence to daily sleep hygiene education, including completion of brief educational sessions delivered by research staff. Adherence reflects the feasibility of implementing behavioral components in a busy inpatient trauma environment.
  Adherence will be summarized descriptively as the proportion of days on which sleep hygiene education was completed. Percentages and confidence intervals will be reported.
Actigraphy Wear-Time Compliance | Throughout the study (upto 7 days of hospital stay)
  Assesses the proportion of hospitalization hours during which the ActiGraph GT3X-BT device records valid data. This measure assesses the feasibility and tolerability of continuous wrist-worn actigraphy in patients with orthopedic trauma.
  Wear-time compliance will be calculated as the percentage of total hospitalization hours with valid actigraphy data. Descriptive statistics (means, SDs, ranges) will be reported.
Retention Through Discharge | Throughout the study (upto 7 days of hospital stay)
  Assesses the proportion of enrolled participants who complete all study procedures through hospital discharge without withdrawal or protocol discontinuation.
  Retention will be summarized as the percentage of participants completing the study through discharge. Proportions and 95% confidence intervals will be reported.
Adverse Events Related to Study Interventions | Throughout the study (upto 7 days of hospital stay)
  Incidence of medication-related side effects (e.g., dizziness, drowsiness, complex sleep behaviors), melatonin intolerance, or actigraphy-related discomfort.
  Adverse events will be summarized using frequencies and proportions. Between-group comparisons may use Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Mara Schenker, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
The study team will share all non-protected data upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon completion of the study.
Access Criteria: Reaching out to the PI.